CLINICAL TRIAL: NCT05886829
Title: A Multicentric, Randomized, Double-Blind, Comparative, Prospective, Placebo-controlled, Phase-II/III Clinical Trial (ACCROS-III)
Brief Title: Chlorpheniramine Nasal Spray to Accelerate COVID-19 Clinical Recovery in an Outpatient Setting: ACCROS-III
Acronym: ACCROS-III
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Dr. Ferrer BioPharma (Industry)
Collaborators: Hospital CEMESA Cortés, San Pedro Sula, Honduras (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DFB-006
Record Dates: First submitted 2023-06-01; First posted 2023-06-02 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-06

CONDITIONS: COVID-19; Symptoms and Signs; COVID-19 Pandemic; Coronavirus Disease 2019; Coronavirus Infections
MeSH Terms: conditions — COVID-19; Signs and Symptoms; Coronavirus Infections | interventions — Chlorpheniramine; Nasal Sprays

STUDY DESIGN:
Intervention Model Description: This is a multi-center, Phase 2/3 Study to evaluate the efficacy and safety of nasally administered CPM in subjects with symptomatic COVID-19 with a positive PCR test.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Chlorpheniramine Malate (0.4%) Nasal Spray (Active Comparator): Chlorpheniramine Malate (0.4%) Nasal Spray
  Interventions: Combination Product: Chlorpheniramine Maleate 0.4% Nasal Spray
- Placebo Nasal Spray (Placebo Comparator): Placebo Nasal Spray
  Interventions: Combination Product: Placebo

INTERVENTIONS:
Combination Product: Chlorpheniramine Maleate 0.4% Nasal Spray — Chlorpheniramine Maleate 0.4% Nasal Spray
  Other Names: ClorNasal; ClorNovir
  Arms: Chlorpheniramine Malate (0.4%) Nasal Spray
Combination Product: Placebo — Placebo nasal spray
  Arms: Placebo Nasal Spray

SUMMARY:
The goal of this clinical trial is to examine the effectiveness of intranasal-administered Chlorpheniramine Maleate in COVID-19-positive participants as part of early treatment for COVID-19. The main questions it aims to answer are:

* To assess the efficacy of nasal spray with Chlorpheniramine (0.4%) for improving clinical recovery in COVID-19 patients.
* To assess the efficacy, safety, and tolerability of nasal spray with Chlorpheniramine (0.4%) as an adjunct to the standard of care in reducing hospitalizations and improving clinical recovery in adult patients with mild COVID-19.

DETAILED DESCRIPTION:
The main goal of the present study is to examine the effectiveness of CPM intranasal spray as part of early treatment for COVID-19. The study will test the hypothesis that intranasal CPM would accelerate clinical recovery, particularly the alleviation of sensory symptoms and URS, in patients with COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients between 18 and 65 years (both inclusive)
* Patients with positive RT-PCR test for SARS-CoV-2 in nasopharyngeal or oropharyngeal swabs (sample collected or proof of positive test ≤3 days before randomization)
* Patients with mild COVID-19 have the following symptoms and signs prior to randomization (≤ 3days)
* Upper respiratory tract symptoms (&/or fever) without shortness of breath or hypoxia. (SpO2 > 94 %)
* Willingness to sign written informed consent document

Exclusion Criteria:

* < 18 years of age
* Hospitalized patients
* Subject with known allergy or hypersensitivity to the components of the formulation.
* Patients receiving therapy with Monoamine oxidase inhibitors (MAOIs): rasagline, selegiline, isocarbonboxasid, phenelzine, tranylcypromine.
* Patients with narrow-angle glaucoma
* urinary retention
* Sleep Apnea
* History of immunodeficiency or receiving immunosuppressive therapy.
* Patients with acute exacerbation of severe comorbidities such as chronic obstructive pulmonary disease (COPD), class 3 and 4 heart failure diagnosed according to the criteria of the New York Heart Failure Association (NYHA), or diseases with severe oxygenation problems
* Any Surgical procedure in the past 12 weeks
* Unable to make informed consent or refuse or renounce adherence to standard treatment protocols.
* Any significant illness or drugs that could interfere with study parameters
* Any other condition based on the investigator's clinical judgment does not justify the patient's participation in the study.
* Participation in another clinical trial within the past 30 days
* Clinically significant arrhythmia or symptomatic cardiac conditions including but not limited to QT elongation
* QT interval less than 300 ms or more than 500 ms for both men and women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2022-07-27 (Actual); Primary Completion 2023-01-19 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Daily symptoms score (DSS) | Baseline through day 7
  Change from baseline daily symptoms score (DSS) to day 7
  The DSS is an instrument comprised of a four-point severity rating scale ranging from 0 to 3.
  0 = no symptoms
  1. = mild symptoms
  2. = moderate symptoms
  3. = severe symptoms.
Visual Analog Scale (VAS) | Baseline through day 7
  Change from baseline visual analog scale (VAS) to day 7
  The VAS is a quantitative method that evaluates the severity of symptoms on a scale of 1-10 (no signs to worst symptoms). A 10 cm line is used to grade the severity of symptoms from "no symptoms" (0 cm) to "the highest level of symptoms" (10 cm).

SECONDARY OUTCOMES:
Hospitalization | Baseline through Day 28
  The proportion of Hospitalizations
Mortality | Baseline through Day 28
  Rate of mortality
The proportion of subjects reporting olfactory function | Baseline through Day 7
  Olfactory function reported on a four-point severity rating scale ranging from 0 to 3.
  0-normal
  1. slightly damaged
  2. moderately damaged
  3. away
The proportion of subjects reporting the presence of upper respiratory symptoms | Baseline through Day 7
  The proportion of subjects reporting the presence of upper respiratory symptoms (anosmia, ageusia, cough, and nasal congestion) using a yes or no scale.
  Yes- Present No- No symptoms present

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital CEMESA, Cortés, San Pedro Sula, Honduras

IPD SHARING:
Plan to Share IPD: Undecided